CLINICAL TRIAL: NCT05387746
Title: Caring Science, Mindful Practice™ and Reiki: Integrative Self-care Approaches to Promote Interprofessional Healthcare Provider Wellbeing
Brief Title: Integrative Self-care Approaches for HCP Wellbeing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Weil Foundation (Unknown)
Responsible Party: Principal Investigator, Linda Kim, Research Scientist II, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00002087
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Burnout, Professional
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Caring Science, Mindful Practice and Reiki Training (Other)
  Interventions: Behavioral: Caring Science, Mindful Practice and Reiki Training

INTERVENTIONS:
Behavioral: Caring Science, Mindful Practice and Reiki Training — Participants will complete a) 4 week internet-based course on Caring Science Mindful Practice and b) 12 hour Reiki training. The participants will also complete online post-training survey with the same questions included in pre-training survey.

SUMMARY:
The purpose of this pilot study is to assess the impact of a hospital-based integrative self-care program (e.g., a. Reiki and b. Caring Science and Mindful Practice [CSMP] course) for interprofessional staff including nurses, physicians and/or medical residents, physical therapists, as well as other healthcare providers on their wellbeing.

DETAILED DESCRIPTION:
The primary research procedures are:

* Participants will complete an online pre-training survey via REDCap, including a demographic questionnaire, and questions related to Physical Function, Depression, Anxiety, Fatigue, Sleep Disturbance, Social Roles/Activities, Resilience, Burnout, COVID-19 Experience, Caring Science, and Reiki Knowledge and Application.
* Participants will participate in the 4-week (virtual) CSMP and (in-person) Reiki Training course.
* Participants will complete the online post-training survey with the same questions included in the pre-training survey.
* Data analysis will be conducted by the research team using descriptive statistics, bivariate analysis, and multivariate linear/logistic regression analysis to assess for relationships between the Reiki and CSMP training and HCP wellbeing.

The research team will enroll up to 20 participants comprising of interprofessional staff including nurses, physicians and/or medical residents, physical therapists, as well as other healthcare providers.

All parts of the protocol will be conducted at CSMC.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare provider must:

  * Be 18 years or older
  * Be full-time employee of a CSMC hospital/clinic
  * MDs/DOs must have admitting privileges to a hospital and/or have private practice/ or be a current medical resident enrolled in a Cedars Sinai Medical Residency Program
  * Provide direct patient care in hospital and/or clinic
  * Consent to participating in the study

Exclusion Criteria:

* Healthcare provider who do not meet all the inclusion criteria and/or reports:

  * They do not provide direct patient care
  * Do not consent to participating in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-08-18 (Actual); Study Completion 2024-08-18 (Actual)

PRIMARY OUTCOMES:
Changes in perception of wellbeing | baseline, 30 days post, and 60 days post-training
  PROMIS® is a publicly available, highly reliable, precise measure of patient-reported health status for physical, mental, and social well-being. Maslach Burnout Inventory covers 3 areas: Emotional Exhaustion, Depersonalization, and low sense of Personal Accomplishment. The investigator chose two items from the MBI as a previous study has shown that relative to the full MBI, single-item measures of emotional exhaustion and depersonalization exhibit strong and consistent associations with key outcomes in various HCWs. Connor-Davidson Resilience Scale is a brief, two-item self-rated measure of resilience, which has shown to have internal consistency, test-retest reliability, convergent validity, and divergent validity as well as significant correlation with the full scale. The investigator will also collect information including demographics, COVID-19 experiences, and knowledge/application of CSMP and Reiki using generic questionnaires that have not been validated.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Kim, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No